CLINICAL TRIAL: NCT00799097
Title: Determinants of Surgical Outcomes in Chronic Sinusitis
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Timothy L. Smith, MD, MPH, Oregon Health & Science University
Other Study IDs: R01 DC0005805; R01DC005805 (NIH)
Record Dates: First submitted 2008-11-26; First posted 2008-11-27 (Estimated); Last update posted 2010-05-20 (Estimated); Status verified 2008-11

CONDITIONS: Chronic Rhinosinusitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Endoscopic Sinus Surgery: Subjects who have failed maximum medical management and have elected for endoscopic sinus surgery

SUMMARY:
Chronic rhinosinusitis (CRS) is a common health condition in the United States resulting in more than 200,000 surgical procedures annually. The field of rhinology has had two major advances which the investigators believe make more accurate prediction of postoperative outcome possible thereby offering the potential of reducing the frequency of unsuccessful surgical procedures. The first advance is the development of validated disease-specific quality of life instruments for measuring outcome of CRS management. The major medical societies now recognize disease-specific quality of life as the gold standard for assessing outcomes in this disease and for the purposes of this study, the investigators define surgical outcome as change in disease-specific quality of life (QOL). The second advance is the better understanding of the pathological process resulting in CRS. The previous construct defined this disease as anatomic obstruction of the sinuses and their secretions. This was thought to be best measured by CT scan which has been the main method of attempting to select the best candidates for surgery.

The investigators hypothesize that utilizing this new conceptual framework, the investigators can better predict surgical outcomes. The investigators will examine several preoperative factors and their relationship to surgical outcome. The factors to be examined include measures of the pathophysiological components of inflammation and anatomic obstruction as well as preoperative extent of disease as measured by preoperative disease-specific quality of life. The investigators hypothesize that these factors provide complimentary information that may be variably expressed in individual CRS patients. Therefore, the investigators hypothesize that a novel integration of multiple preoperative factors will form a useful predictive model of surgical outcome. Finally this prospective study provides the opportunity to add to the field by identifying potentially novel risk factors and comorbidities as well as study secondary outcomes of sinus surgery including olfactory function and general health related quality of life in a systematic manner.

DETAILED DESCRIPTION:
A cohort of 500+ patients with CRS undergoing sinus surgery at three centers will be prospectively enrolled. Patient demographics, comorbidity data, objective testing, and QOL evaluation will occur preoperatively and outcomes (QOL and olfactory testing) will be measured 6, 12, and 18 months postoperatively. Determinants of change in QOL will be analyzed by univariate and multivariate methods including construction of a multivariate predictive model.

This proposal focuses on patients undergoing surgical intervention for the management of CRS. The findings can potentially be applied to the 200,000 patients annually undergoing sinus surgery and in working toward the long-term goal of developing a comprehensive system for measuring extent of disease so that disease severity and treatment response can be rigorously quantified in the 30 million patients with CRS.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years and older) (see Inclusion of Children)
* CRS by Rhinosinusitis Task Force criteria
* Symptoms persisting following standard medical management as outlined in the Research Design and Methods.
* Elect sinus surgery and give informed consent.
* Patient must be able to travel to the Institution of enrollment for evaluation, treatment, and follow up.
* Patient must be able to complete a questionnaire with the assistance of the Study Coordinator and be able to cooperate with endoscopy, olfactory and CT studies.
* Patient (if White) selected by randomized enrollment technique

Exclusion Criteria:

* Unable to complete questionnaires or cooperate with studies
* Children (<18 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The multi-institutional study population consists of adult (>17 years) patients who have had a diagnosis of chronic rhinosinusitis, have failed maximum medical management,and have elected for endoscopic sinus surgery as their next treatment option.
Sampling Method: Non-Probability Sample
Enrollment: 516 (Actual)
Dates: Start 2004-07; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Disease specific quality of life | Preoperatively, 6 months, 12 months, 18 months

SECONDARY OUTCOMES:
General quality of life | Preoperatively, 6 months, 12 months, 18 months
Olfactory function | Preoperatively, 6 months, 12 months, 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Timothy L Smith, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Stewart MG, Smith TL. Objective versus subjective outcomes assessment in rhinology. Am J Rhinol. 2005 Sep-Oct;19(5):529-35. PMID 16270610
- [Background] Martin TJ, Yauck JS, Smith TL. Patients undergoing sinus surgery: constructing a demographic profile. Laryngoscope. 2006 Jul;116(7):1185-91. doi: 10.1097/01.mlg.0000224506.42567.6e. PMID 16826058
- [Background] Chester AC, Sindwani R, Smith TL, Bhattacharyya N. Fatigue improvement following endoscopic sinus surgery: a systematic review and meta-analysis. Laryngoscope. 2008 Apr;118(4):730-9. doi: 10.1097/MLG.0b013e318161e57b. PMID 18216743
- [Result] Smith TL, Mendolia-Loffredo S, Loehrl TA, Sparapani R, Laud PW, Nattinger AB. Predictive factors and outcomes in endoscopic sinus surgery for chronic rhinosinusitis. Laryngoscope. 2005 Dec;115(12):2199-205. doi: 10.1097/01.mlg.0000182825.82910.80. PMID 16369166
- [Result] Mendolia-Loffredo S, Laud PW, Sparapani R, Loehrl TA, Smith TL. Sex differences in outcomes of sinus surgery. Laryngoscope. 2006 Jul;116(7):1199-203. doi: 10.1097/01.mlg.0000224575.12945.90. PMID 16826060
- [Result] Poetker DM, Mendolia-Loffredo S, Smith TL. Outcomes of endoscopic sinus surgery for chronic rhinosinusitis associated with sinonasal polyposis. Am J Rhinol. 2007 Jan-Feb;21(1):84-8. doi: 10.2500/ajr.2007.21.2978. PMID 17283567
- [Result] Reh DD, Mace J, Robinson JL, Smith TL. Impact of age on presentation of chronic rhinosinusitis and outcomes of endoscopic sinus surgery. Am J Rhinol. 2007 Mar-Apr;21(2):207-13. doi: 10.2500/ajr.2007.21.3005. PMID 17424882
- [Result] Robinson JL, Griest S, James KE, Smith TL. Impact of aspirin intolerance on outcomes of sinus surgery. Laryngoscope. 2007 May;117(5):825-30. doi: 10.1097/MLG.0b013e3180333121. PMID 17473677
- [Result] Litvack JR, Griest S, James KE, Smith TL. Endoscopic and quality-of-life outcomes after revision endoscopic sinus surgery. Laryngoscope. 2007 Dec;117(12):2233-8. doi: 10.1097/MLG.0b013e31814539e8. PMID 17891047
- [Result] Mace J, Michael YL, Carlson NE, Litvack JR, Smith TL. Effects of depression on quality of life improvement after endoscopic sinus surgery. Laryngoscope. 2008 Mar;118(3):528-34. doi: 10.1097/MLG.0b013e31815d74bb. PMID 18043488
- [Result] Poetker DM, Litvack JR, Mace JC, Smith TL. Recurrent acute rhinosinusitis: presentation and outcomes of sinus surgery. Am J Rhinol. 2008 May-Jun;22(3):329-33. doi: 10.2500/ajr.2008.22.3177. PMID 18588769
- [Result] Soler ZM, Mace J, Smith TL. Symptom-based presentation of chronic rhinosinusitis and symptom-specific outcomes after endoscopic sinus surgery. Am J Rhinol. 2008 May-Jun;22(3):297-301. doi: 10.2500/ajr.2008.22.3172. PMID 18588763
- [Result] Sautter NB, Mace J, Chester AC, Smith TL. The effects of endoscopic sinus surgery on level of fatigue in patients with chronic rhinosinusitis. Am J Rhinol. 2008 Jul-Aug;22(4):420-6. doi: 10.2500/ajr.2008.22.3196. PMID 18702910
- [Result] Soler ZM, Mace J, Smith TL. Fibromyalgia and chronic rhinosinusitis: outcomes after endoscopic sinus surgery. Am J Rhinol. 2008 Jul-Aug;22(4):427-32. doi: 10.2500/ajr.2008.22.3198. PMID 18702911
- [Derived] Soler ZM, Hyer JM, Rudmik L, Ramakrishnan V, Smith TL, Schlosser RJ. Cluster analysis and prediction of treatment outcomes for chronic rhinosinusitis. J Allergy Clin Immunol. 2016 Apr;137(4):1054-1062. doi: 10.1016/j.jaci.2015.11.019. Epub 2016 Jan 22. PMID 26806047
- [Derived] Rudmik L, Mace J, Soler ZM, Smith TL. Long-term utility outcomes in patients undergoing endoscopic sinus surgery. Laryngoscope. 2014 Jan;124(1):19-23. doi: 10.1002/lary.24135. Epub 2013 May 13. PMID 23670699
- [Derived] Soler ZM, Mace JC, Litvack JR, Smith TL. Chronic rhinosinusitis, race, and ethnicity. Am J Rhinol Allergy. 2012 Mar-Apr;26(2):110-6. doi: 10.2500/ajra.2012.26.3741. PMID 22487286
- [Derived] Rudmik L, Mace J, Ferguson BJ, Smith TL. Concurrent septoplasty during endoscopic sinus surgery for chronic rhinosinusitis: does it confound outcomes assessment? Laryngoscope. 2011 Dec;121(12):2679-83. doi: 10.1002/lary.22361. Epub 2011 Oct 27. PMID 22034233
- [Derived] Soler ZM, Wittenberg E, Schlosser RJ, Mace JC, Smith TL. Health state utility values in patients undergoing endoscopic sinus surgery. Laryngoscope. 2011 Dec;121(12):2672-8. doi: 10.1002/lary.21847. Epub 2011 Oct 27. PMID 22034223
- [Derived] Bhandarkar ND, Mace JC, Smith TL. The impact of osteitis on disease severity measures and quality of life outcomes in chronic rhinosinusitis. Int Forum Allergy Rhinol. 2011 Sep-Oct;1(5):372-8. doi: 10.1002/alr.20068. PMID 22028948
- [Derived] Rudmik L, Mace JC, Smith TL. Smoking and endoscopic sinus surgery: does smoking volume contribute to clinical outcome. Int Forum Allergy Rhinol. 2011 May-Jun;1(3):145-52. doi: 10.1002/alr.20045. PMID 21731825
- [Derived] Rudmik L, Mace J, Smith T. Low-stage computed tomography chronic rhinosinusitis: what is the role of endoscopic sinus surgery? Laryngoscope. 2011 Feb;121(2):417-21. doi: 10.1002/lary.21382. PMID 21271599
- [Derived] Soler ZM, Sauer DA, Mace JC, Smith TL. Ethmoid histopathology does not predict olfactory outcomes after endoscopic sinus surgery. Am J Rhinol Allergy. 2010 Jul-Aug;24(4):281-5. doi: 10.2500/ajra.2010.24.3477. PMID 20819467
- [Derived] Khalid AN, Mace JC, Smith TL. Outcomes of sinus surgery in ambulatory patients with immune dysfunction. Am J Rhinol Allergy. 2010 May-Jun;24(3):230-3. doi: 10.2500/ajra.2010.24.3464. PMID 20537292
- [Derived] Mace JC, Michael YL, Carlson NE, Litvack JR, Smith TL. Correlations between endoscopy score and quality of life changes after sinus surgery. Arch Otolaryngol Head Neck Surg. 2010 Apr;136(4):340-6. doi: 10.1001/archoto.2010.34. PMID 20403849
- [Derived] Soler ZM, Hwang PH, Mace J, Smith TL. Outcomes after middle turbinate resection: revisiting a controversial topic. Laryngoscope. 2010 Apr;120(4):832-7. doi: 10.1002/lary.20812. PMID 20232413
- [Derived] Soler ZM, Sauer D, Mace J, Smith TL. Impact of mucosal eosinophilia and nasal polyposis on quality-of-life outcomes after sinus surgery. Otolaryngol Head Neck Surg. 2010 Jan;142(1):64-71. doi: 10.1016/j.otohns.2009.10.005. Epub 2009 Nov 22. PMID 20096225
- [Derived] Smith TL, Litvack JR, Hwang PH, Loehrl TA, Mace JC, Fong KJ, James KE. Determinants of outcomes of sinus surgery: a multi-institutional prospective cohort study. Otolaryngol Head Neck Surg. 2010 Jan;142(1):55-63. doi: 10.1016/j.otohns.2009.10.009. PMID 20096224